CLINICAL TRIAL: NCT06238492
Title: Intervening Quickly: A Pilot RCT to Improve Cognitive Processing Speed in Acute SCI
Brief Title: A Pilot RCT to Improve Cognitive Processing Speed in Acute SCI
Acronym: SCI-IQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Craig Hospital (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Erica Weber, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-1210-23
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries; Cognitive Dysfunction; Cognitive Impairment; Acute Spinal Cord Injury
Keywords: processing speed
MeSH Terms: conditions — Spinal Cord Injuries; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): pre-specified computer tasks using an Internet-based cognitive training portal, to be completed 3x per week for 60 minutes each session for 12 weeks total
  Interventions: Behavioral: game-like computerized activities
- Placebo Control (Placebo Comparator): pre-specified computer tasks using an Internet-based cognitive training portal, to be completed 3x per week for 60 minutes each session for 12 weeks total
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: game-like computerized activities — Experimental
  Arms: Experimental
Behavioral: Placebo — game-like computerized activities
  Arms: Placebo Control

SUMMARY:
This study seeks conduct a pilot study to test whether a cognitive training program can improve processing speed abilities in individuals with acute traumatic spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) newly affects approximately 18,000 persons in the US per year. Decades of research have focused on the physical limitations associated with SCI, as well as therapies for addressing these physical problems. However, it is becoming better acknowledged that many individuals experience significant problems with their cognitive abilities, such as attention, memory, and the time it takes them to process information. Research has shown that people who have cognitive difficulties, compared to those with a purely physical disability, are less likely to be employed, engage in fewer social and work-related activities, have greater difficulties carrying out routine household tasks, and are at higher risk for mental illness. If cognitive issues arise after an SCI, it is more likely that a person would have a more challenging time adapting the many lifestyle changes brought about by their injury, would benefit less from their rehabilitation program, and have more difficulty rejoining the workforce. As it stands, cognitive assessment or rehabilitation is not part of the standard of care for individuals after their SCI because of the relative lack of research in this area. This study seeks conduct a multisite pilot study to test whether a cognitive training program can improve processing speed abilities in individuals shortly after they experience their SCI, with the hopes that this early intervention will improve the trajectory of their overall health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* 18-59 years old
* recent traumatic SCI (approximately 6 months post-injury)

Exclusion Criteria:

* no other significant neurological, psychiatric or substance use history
* no significantly impairing visual disturbance

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-29 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Useful Field of View (UFOV) | baseline to immediate post-treatment (week 13) and long-term follow-up (week 25)
  computerized processing speed task
Letter & Pattern Comparison (LPC) | baseline to immediate post-treatment (week 13) and long-term follow-up (week 25)
  processing speed task, using both letter and pattern strings
Symbol Digit Modalities Test (SDMT) | baseline to immediate post-treatment (week 13) and long-term follow-up (week 25)
  processing speed task, matching numbers to symbols using a key

SECONDARY OUTCOMES:
Spinal Cord Injury Quality of Life scales | baseline to immediate post-treatment (week 13) and long-term follow-up (week 25)
  self-reported instruments of quality of life after SCI

CONTACTS AND LOCATIONS:
Overall Officials: Erica Weber, PhD, Principal Investigator — Kessler Foundation
Locations (3):
- United States (3):
  - Craig Hospital, Englewood, Colorado
  - Kessler Foundation, East Hanover, New Jersey
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No